CLINICAL TRIAL: NCT05774535
Title: Prospective, Observational Study on the Investigation of the Carotid Intima-media Thickness in Patients Undergoing Thyroid Surgery
Brief Title: Prospective, Observational Study on the Carotid Intima-media Thickness in Patients Undergoing Thyroid Surgery
Acronym: TIROVASC
Status: Withdrawn | Type: Observational
Why Stopped: No enrollment
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 34C211
Record Dates: First submitted 2023-02-22; First posted 2023-03-17 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Plummer Disease; Multinodular Goiter; Graves Disease; Hyperthyroidism; Euthyroid Goiter; Thyroid Cancer; Basedow Disease
Keywords: carotid intima-media thickness; cardiovascular disease; thyroid disease; carotid artery
MeSH Terms: conditions — Graves Disease; Hyperthyroidism; Euthyroid Goiter; Thyroid Neoplasms; Cardiovascular Diseases; Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Patients who will undergo thyroidectomy
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Experimental — Patients will undergo thyroidectomy according to the guidelines American Thyroid Association (ATA), Randolph.
  The following assessments will be performed within 10 days before the thyroidectomy procedure:
  * informed consent;
  * personal data and medical records;
  * registration of medical therapy and post-procedural pharmacological protocol
  * surgical check;
  * supra-aortic trunks EchocolorDoppler;
  * pre-procedural blood sampling.
  The following assessments will be performed after 30 days, 6 months and 12 months from the thyroidectomy procedure:
  * surgical checks;
  * registration of drug therapy;
  * recording of all adverse events that occurred during hospitalization
  * supra-aortic trunks EchocolorDoppler and cIMT measurement;
  * blood sampling.

SUMMARY:
The evaluation of carotid intima-media thickness (cIMT) has become a possible predictor of the future risk of cardiovascular diseases (CVD). Evidence to date shows that cIMT augmentation is correlated with the extent of atherosclerosis in the coronary arteries and with other risk factors for CVD. More recently, several studies have evaluated the association of cIMT with stroke, to determine whether this measure can also predict future cardiovascular events.

Although the published evidence is scarce and fragmentary, the cIMT retains an increasingly interesting role as a marker of atherosclerotic pathology.

The purpose of the study is to analyze cIMT in patients undergoing thyroidectomy to evaluate a possible correlation between the cIMT variation after the procedure and the cause of the thyroid disease, the levels of thyroid hormones, and the lipid or other markers of atherosclerosis levels.

The primary endpoint will be the variation of the measure of the cIMT before and after surgery.

Secondary endpoints will be:

* major cardiovascular adverse events (death, major stroke, minor stroke, transient ischemic attack) in the short-term period (≤30 days after the procedure);
* major cardiovascular adverse events (death, major stroke, minor stroke, transient ischemic attack) in the long-term period (>30 days after the procedure);
* the technical success of the procedure;
* the rate of postoperative complications. To date, there are no data that differentiate patients based on the causes of thyroid disease. The results of the present study will allow for correlating the variation of the cIMT to the causes of thyroid disease, the levels of thyroid hormones, and the levels of lipid and other markers of atherosclerosis.

Results from the present study may provide insights into possible areas of quality improvement. It may also influence the economic impact associated with carotid revascularization techniques, in terms of hospital charges and discharges to skilled nursing and rehabilitation facilities.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thyroidectomy according to the American Thyroid Association (ATA), International neural monitoring study group guideline (INMSG), Italian Society of Endocrine Surgery (SIUEC);
* subjects who have read and signed the informed consent;
* subjects who undertake to undergo the instrumental examinations and visits necessary for the study during the follow-up;
* >18 years of age.

Exclusion Criteria:

* occlusion or stenosis of at least one carotid artery, with plaque > 30%;
* exposure to ionizing radiation;
* previous neck, carotid (endarterectomy or stenting) and/or thyroid surgery;
* clinical conditions that preclude proper follow-up;
* HIV, dialysis therapy and all clinical conditions with increased cIMT;
* uncontrolled dyslipidemia;
* pregnant and breastfeeding women;
* terminal patients.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the potential eligible candidates will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Carotid Intima-Media Thickness (cIMT) | Baseline (10 days before the surgery), 30 days, 6 months and 12 months after the surgery
  cIMT is a measurement of the thickness of tunica intima and tunica media, the innermost two layers of the wall of an artery. The measurement is made by external ultrasound according to the recommendation of the Joint Carotid Intima-Media Thickness and Plaque Area Measurement in Ultrasound for Cardiovascular/Stroke Risk Monitoring.

SECONDARY OUTCOMES:
Cumulative incidence of adverse events during periprocedural period | Within 30 days after the surgery
  Incidence of death, major stroke, minor stroke, transient ischemic attack
Cumulative incidence of adverse events during postprocedural period | Between 30 days after the surgery and 12 months after surgery
  Incidence of death, major stroke, minor stroke, transient ischemic attack
Change from baseline in lipid profile | Baseline (10 days before the surgery), 30 days, 6 months and 12 months after the surgery
  Total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano , IRCCS, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes